CLINICAL TRIAL: NCT02298998
Title: Surveillance for Low and Low-Intermediate Risk Non-muscle Invasive Bladder Cancer: A Pilot Study
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC20130177H
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — After participant signs the consent form, research staff may ask participant to provide a urine sample at each study visit for research purposes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention: The intervention group refers to surveillance based on the EAU guidelines.
  Interventions: Other: Intervention
- Control: The control group refers to surveillance based on the AUA guidelines.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Patients randomized into the intervention group will follow the European Urologic Association (EAU) surveillance guidelines for cystoscopy follow-ups during bladder cancer surveillance.
  Other Names: EAU surveillance
  Groups: Intervention
Other: Control — Patients randomized into the control group will follow the American Urologic Association (AUA) surveillance guidelines using cystoscopy ever 3 months for the first two years, and then every 6 months for 2 years.
  Other Names: AUA Surveillance
  Groups: Control

SUMMARY:
This is a two-arm, randomized-controlled pilot study with 2 year duration. The "intervention" refers to surveillance based on the European Association of Urology (EAU) guidelines and the "control" refers to surveillance based on the American Urological Association (AUA) guidelines.

DETAILED DESCRIPTION:
This is a two-arm, randomized-controlled pilot study with 2 year duration. The "intervention" refers to surveillance based on the EAU guidelines and the "control" refers to surveillance based on the AUA guidelines.

Research methods: Participants who presents with non-muscle invasive bladder cancer and meets the inclusion/exclusion criteria will be given an option to participate in the study. Participants will be enrolled at the Urology Clinics at the University of Texas Health Science Center San Antonio (UTHSCSA) Medical Arts and Research Center (MARC) and South Texas Veterans Health Care System (STVHCS). Non-local site include the University of Texas Southwestern Medical Center (UTSW). The research procedures consist of urine collection, cystoscopy, and patient satisfaction and cost questionnaires. The evaluation will be done by the tumor recurrence and progression of the disease. At various time points throughout the study, urine may be obtained from the patient and banked in the Genitourinary (GU) Tissue Bank. Subjects asked to provide a urine sample(s) will be asked to sign a separate informed consent. The urine is de-identified in the lab per the Health Insurance Portability and Accountability Act (HIPAA) protocol GU Tissue Bank Institutional Review Board (IRB) # 20050234H). Patients will undergo cystoscopy in clinic (standard of care). In the intervention arm, patient surveillance cystoscopy will be performed at 3, 12 months and again at 24 months following the diagnosis of bladder cancer. Patients randomized to the control arm, will undergo surveillance cystoscopy every 3 months for 2 years following the diagnosis of bladder cancer. Because use of cytology is variable among the participating urologist, the utilization of cytology will be at the treating urologist's discretion as per usual standard care. Study duration will be 2 years from most recent biopsy. Patients will be placed on the surveillance schedule based on the length of time from their last tumor.

ELIGIBILITY:
Inclusion Criteria:

* Must have non-muscle invasive low-grade, papillary (Ta) bladder cancer.
* Must have a negative cystoscopy following most recent biopsy.
* Must be able to give informed consent.
* Must be age 18 or older.
* Must be at low- or low-intermediate risk for disease recurrence and progression according to the EAU guidelines.

Exclusion Criteria:

* Have a history of invasive (>=T1) bladder cancer.
* Have a history of carcinoma-in-situ (CIS).
* Unable to give informed consent.
* < 18 or younger.
* Variant histology (micropapillary, nested variant, non-urothelial cell carcinoma elements).
* Had a surveillance cystoscopy following most recent biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of low or low-intermediate risk non-muscle invasive bladder cancer. They are being followed with periodic examinations of their bladder as a means for cancer surveillance.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-03; Primary Completion 2021-05-28 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate feasibility of study recruitment and retention in order to help plan for subsequent phase III study. | 2 years
Develop methods for assessing patient satisfaction and costs associated with cystoscopy during bladder cancer surveillance. | 2 years

SECONDARY OUTCOMES:
Capture preliminary data regarding number of procedures and direct and indirect cost differences between study arms. | 2 years
Compare proportion of patients experiencing disease progression and recurrence at 2 years following most recent biopsy under two different surveillance approaches. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center, San Antonio, Texas, United States